CLINICAL TRIAL: NCT06184048
Title: Validation of a Low-cost Platelet-Rich Plasma (PRP)
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Daniel Cushman, Principle Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00159071
Record Dates: First submitted 2022-10-31; First posted 2023-12-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Platelet-Rich Plasma (PRP); Knee Osteoarthritis (OA)
Keywords: Platelet-Rich Plasma; PRP; Neutrophil-poor PRP
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Recruitment will take place at the University of Utah Orthopedic Center by physician and study study staff members EMR chart review prior to patient visits.
  The investigator plans to recruit a total of 30 participants to this project over a 24 month period of time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Directly Address Two Concerns - Proper Reporting of PRP Composition and Greatly Decreasing Cost (Other): As socioeconomic inequity directly relates to disability related to knee Osteoarthritis (OA), limiting the cost of treatment is of the utmost importance to ensure appropriate delivery of care to all patients. As PRP is currently not covered by the vast majority of public and private payors, patients are required to pay for the injections out of pocket, with an average cost of $714 per injection (as high as $2,092). Furthermore, research studies relating to PRP are often expensive due to the cost of the traditional method of extracting PRP, generally with commercial kits, and thus limited in scope. The investigators have developed and implemented a low-cost PRP (LC-PRP) preparation technique and have safely performed the injections on hundreds of patients with knee OA.
  Interventions: Procedure: Intra-Articular knee injection of LC-PRP

INTERVENTIONS:
Procedure: Intra-Articular knee injection of LC-PRP — Blood Collection 45mL, Processed Neutrophil-Poor PRP, 2 Injections at day 0 and 3 weeks.

SUMMARY:
Knee osteoarthritis is an extremely common and debilitating condition, more common in women, with an estimated global prevalence of 16%, and as high as 50% by the age of 80. Current management of knee osteoarthritis (OA) revolves around conservative treatments- biomechanical interventions, intra-articular injections, exercise, self-management and education, oral or topical medications, strength training, and weight management - or surgical management. For injection therapies, corticosteroids remain the standard of care; approximately 84% of sports medicine physicians perform these knee injections at least monthly, reporting a median range of 11-20 injections per month. Multiple detrimental effects of corticosteroid injections are well-known, including alterations of the hypothalamic-pituitary-adrenal axis, blood glucose levels, bone turnover, inflammatory response, blood pressure, and psychologic well-being. Thus, alternative therapies are of the utmost importance.

Platelet-Rich Plasma (PRP) is an injectable preparation of a patient's blood that can be used for numerous conditions and has received significant attention over the past several years for its potential application for the treatment of pain and functional impairment due to knee OA. Systematic reviews of randomized-controlled trials have demonstrated equivalent-to-superior treatment outcomes associated with the use of intra-articular PRP compared to placebo, hyaluronic acid, and corticosteroid. Furthermore, use of intra-articular PRP is associated with a very low rate of adverse events and is likely safer than injectable corticosteroids. Concerns that have limited a wider use of PRP include two main concerns - an uncertainty regarding the current evidence base due to study-related bias, heterogeneity, and lack of reporting standards; and second, more importantly, the main issue remains high cost.

DETAILED DESCRIPTION:
Study Purposes and Objectives:

The study will directly address two concerns - proper reporting of PRP composition and greatly decreasing cost. As socioeconomic inequity directly relates to disability related to knee Osteoarthritis (OA), limiting the cost of treatment is of the utmost importance to ensure appropriate delivery of care to all patients. As PRP is currently not covered by the vast majority of public and private payors, patients are required to pay for the injections out of pocket, with an average cost of $714 per injection (as high as $2,092). Furthermore, research studies relating to PRP are often expensive due to the cost of the traditional method of extracting PRP, generally with commercial kits, and thus limited in scope. The investigators have developed and implemented a low-cost PRP (LC-PRP) preparation technique and have safely performed the injections on hundreds of patients with knee OA. The cost of this preparation technique is equivalent to the cost of a vial of corticosteroid and it is easy to replicate. In conjunction with Internal Departmental matching funds, this grant will cover the cost of resources to support the study, which will allow for future clinical and research endeavors in this realm.

The primary goal of this study is to validate this easy-to-replicate LC-PRP preparation technique to demonstrate that its composition is equivalent to standard, commercially-available PRP preparation kits. Validation must include data that match the minimum reporting standards for clinical studies evaluating PRP. Once validated, this will allow for a low-cost method to prepare PRP in countless clinical and research realms. Specifically, the investigators will analyze the components of both the whole blood (the subject's blood from which the PRP is extracted) and the PRP itself. Based on extensive pilot data, the platelet yield - the amount of platelets extracted from the patient's whole blood - is equivalent to those seen from expensive, commercially-available kits. Though this study will use neutrophil-poor PRP, this method can just as easily create neutrophil-rich PRP for other future clinical needs.

The investigators secondary goal is to prospectively evaluate pain and functional outcomes in a cohort of patients with knee OA. Based on the investigators pilot data, zero significant adverse events have been reported after treatment of over 1,000 patients with this technique in two separate geographical regions. The investigators have incomplete clinical outcome data, but it preliminarily demonstrates positive outcomes at 3 and 6 months in cohort. The investigators plan on using the results of this validation study to seek external funding for a randomized-controlled trial (RCT) comparing LC-PRP to corticosteroid injection for knee OA.

The investigator's tertiary goal is to conduct a cost-effectiveness analysis of LC-PRP compared to corticosteroid injection from a payor perspective using a computer simulation model. This simulation model, to be performed by Dr. Nelson, will be parameterized using a combination of data from the proposed study and from previously published literature. This model will also be a stepping stone for a cost-effectiveness analysis that will be conducted alongside the aforementioned future RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any adult age with symptomatic Kellgren-Lawrence (K-L) score 1-3 knee OA, based on radiographs within the last six months.
2. Patients must have failed at least six weeks of conventional conservative treatments (such as medication or physical therapy).
3. Patients with bilateral knee OA will only be eligible if both knees fit the criteria; each knee will count separately.

Exclusion Criteria:

1. Recent (last two years) knee surgery,
2. Prior orthobiologic injection(s) into the knee,
3. Known major axial deviation (over 30 degrees)
4. Known thrombocytopenia (platelets under 50,000), thrombocythemia (platelets over 1,000,000), known platelet disorder (ITP, TTP, or Lowe syndrome)
5. Active systemic infection requiring antibiotics, or local infection at the site of injection,
6. Non-ambulatory patients,
7. Patients seeking care with active litigation pending
8. Body mass index (BMI) over 40
9. Injection into the affected joint within the last six months
10. Oral steroids consumed within the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to validate our easy-to replicate LC-PRP preparation technique | 24-Months
  The primary goal of this study is to validate the investigator(s) easy-to-replicate LC-PRP preparation technique to demonstrate that its composition is equivalent to standard, commercially-available PRP preparation kits. The investigators will specifically compare the quantity of platelets derived from their system compared to previously published platelet counts for commercially available PRP preparation kits.

SECONDARY OUTCOMES:
Pain and functional outcomes | 24-Months
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score at 1, 3, 6, and 12 months after the second injection. Lastly, the investigator(s) will be evaluating adverse events for safety purposes.(functional and pain measure)
QOL outcomes | 24-Months
  EQ-5D (EuroQual, quality of life measure) at 1, 3, 6, and 12 months after the second injection. Lastly, the investigator(s) will be evaluating adverse events for safety purposes.
Global impression of change | 24-Months
  Global impression of change at 1, 3, 6, and 12 months after the second injection.
Patient Satisfaction (GPS) | 24-Months
  Global patient satisfaction (GPS) at 1, 3, 6, and 12 months after the second injection.

OTHER OUTCOMES:
Cost-effectiveness | 24-Months
  Cost inputs for this simulation model will consist of intervention and healthcare costs. The current total cost for a corticosteroid injection includes medication, physician fee, facility fee, and supplies. The LC-PRP has a slightly higher supply cost, and a non-existent medication cost. We will be monitoring and recording the amount of time it takes for each task to accurately identify facility- and personnel-related time-costs.
Healthcare utilization | 24-Months
  We will obtain healthcare utilization following the intervention for patients in this study. These will then be combined with unit costs from Medicare to construct direct medical costs from the payer perspective for patients in the LC-PRP arm of our model.
Direct medical costs | 24-Months
  Direct medical costs for patients in the corticosteroid arm of our model will be obtained from the published literature. We will use this model to estimate the expected cost and effectiveness for both strategies and construct an incremental cost-effectiveness ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cushman, MD, Principal Investigator — University of Utah Orthopedic Center
Locations (1):
- University of Utah Orthopedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu J, Duan W, Yu Z, Tao T, Xu J, Ma Q, Zhao L, Guo JJ. Intra-articular injections of platelet-rich plasma decrease pain and improve functional outcomes than sham saline in patients with knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2022 Dec;30(12):4063-4071. doi: 10.1007/s00167-022-06887-7. Epub 2022 Feb 6. PMID 35124707
- [Background] Dai WL, Zhou AG, Zhang H, Zhang J. Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2017 Mar;33(3):659-670.e1. doi: 10.1016/j.arthro.2016.09.024. Epub 2016 Dec 22. PMID 28012636
- [Background] Chu CR, Rodeo S, Bhutani N, Goodrich LR, Huard J, Irrgang J, LaPrade RF, Lattermann C, Lu Y, Mandelbaum B, Mao J, McIntyre L, Mishra A, Muschler GF, Piuzzi NS, Potter H, Spindler K, Tokish JM, Tuan R, Zaslav K, Maloney W. Optimizing Clinical Use of Biologics in Orthopaedic Surgery: Consensus Recommendations From the 2018 AAOS/NIH U-13 Conference. J Am Acad Orthop Surg. 2019 Jan 15;27(2):e50-e63. doi: 10.5435/JAAOS-D-18-00305. PMID 30300216
- [Background] Belk JW, Kraeutler MJ, Houck DA, Goodrich JA, Dragoo JL, McCarty EC. Platelet-Rich Plasma Versus Hyaluronic Acid for Knee Osteoarthritis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Am J Sports Med. 2021 Jan;49(1):249-260. doi: 10.1177/0363546520909397. Epub 2020 Apr 17. PMID 32302218